CLINICAL TRIAL: NCT06880146
Title: Cross-validation of a Predictive Model of Response to Anti-TNF Alpha Based on Oxylipin Response in Rheumatoid Arthritis
Acronym: OPERAVAL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Unité de Nutrition Humaine, INRAE, Centre Auvergne-Rhône Alpes (Unknown); Immunology department, CHU Clermont-Ferrand (Unknown); University of Southampton, Southampton, United Kingdom (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RBHP 2024 TOURNADRE
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid, arthritis; Oxylipin; Cytokin; EULAR response; Polyunsaturated fat
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: Cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cohort (Other): Intervention : blood sample added to the standard blood test at visit Inclusion and Month 6.
  Interventions: Other: Blood sample Truculture

INTERVENTIONS:
Other: Blood sample Truculture — blood sample added to the standard blood test at visit Inclusion and Month 6. This project will use the TruCulture® Whole Blood Stimulation System to assess the Whole Blood Oxylipin Response (WBOR).
  WBOR is the ability of patients to produce oxylipins in response to an immune stimulus. One tube is conditioned with LPS stimulant and a control tube is conditioned with no stimulant (Null).

SUMMARY:
The goal of this clinical trial is to use a blood test to predict whether a participant diagnosed with rheumatoid arthritis will respond to anti-TNF alpha treatment . The main questions it aims to answer is:

Is the predictive model created using oxylipins effective?

Participants starting anti-TNF alpha treatment will have a blood sample taken before starting treatment and 6 months afterwards.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient aged 18 years or older with rheumatoid arthritis according to ACR EULAR 2010 criteria
* Active disease as defined by DAS-28-CRP>3.2
* Naive to targeted biologic or synthetic therapy
* Rheumatologist's decision to start anti-TNFα treatment
* Stable corticosteroid therapy ≤ 10 mg/day
* Patient enrolled in or benefiting from a social security scheme
* Patient who has given written informed consent to participate in the study

Exclusion Criteria:

* Contraindication to biological treatment (cancer or history of cancer)
* Treatment with non-steroidal anti-inflammatory drugs in the 2 weeks prior to enrolment
* Protected persons (pregnant and/or breastfeeding women, persons under guardianship or conservatorship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Whole Blood Oxylipin Response (WBOR) | Month 0
  i.e. the ability of the host's blood cells to produce oxylipins in response to an immune stimulus. A wide range of several dozen pro- and anti-inflammatory oxylipins secreted by stimulated blood cells.
EULAR clinical response | Month 6
  EULAR clinical response (based on change in DAS28 score) assessed after 6 months of anti-TNFα treatment. EULAR non-responders are defined as RA patients who did not achieve a good or moderate EULAR response after 6 months of treatment, discontinued the drug, started a new bDMARD or increased the oral corticosteroid dose to more than 10 mg/d at the second visit.

SECONDARY OUTCOMES:
Performance of the predictive response model | Month 0
  The predictive performance of the model in the validation study is evaluated and compared using a ROC curve (Receiver Operating Characteristic Curve).
Polyunsaturated fat (PUFA) content of blood cells | Month 0
  PUFA content of blood cells (leukocytes, red blood cells and platelets) present in the cell pellet in the Truculture tube.
Polyunsaturated fat (PUFA) content of blood cells | Month 6
  PUFA content of blood cells (leukocytes, red blood cells and platelets) present in the cell pellet in the Truculture tube.
Cytokine response | Month 0
  Large panel of 21 cytokines characteristic of the inflammatory response and lymphocyte polarisation (IL-1β, IFN-α2, IFN-γ, TNF-α, MCP-1 (CCL2), IL-6, IL-8 (CXCL8), IL-10, IL-12p70, IL-17A, IL-18, IL-23, IL-33, IL-5, IL-13, IL-2, IL-9, IL-10, IL-17F, IL-4, IL-22).
Cytokine response | Month 6
  Large panel of 21 cytokines characteristic of the inflammatory response and lymphocyte polarisation (IL-1β, IFN-α2, IFN-γ, TNF-α, MCP-1 (CCL2), IL-6, IL-8 (CXCL8), IL-10, IL-12p70, IL-17A, IL-18, IL-23, IL-33, IL-5, IL-13, IL-2, IL-9, IL-10, IL-17F, IL-4, IL-22).
Whole Blood Oxylipin Response (WBOR) | Month 6
  a wide range of several dozen pro- and anti-inflammatory oxylipins secreted by stimulated blood cells

CONTACTS AND LOCATIONS:
Overall Officials: Anne TOURNADRE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (3):
- France (3):
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - Hopital Cochin, APHP, Paris
  - CHU Saint Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No